CLINICAL TRIAL: NCT04422392
Title: Neoadjuvant PD-1 Antibody Plus Chemotherapy in Resectable Stage IIIA-N2 Non-Small-Cell Lung Cancer: A Randomized Phase II Study
Brief Title: Neoadjuvant PD-1 Antibody Plus Chemotherapy in Resectable Stage IIIA-N2 Non-Small-Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: since the CheckMate816 study is published in NEJM, enrolling patients becomes difficult
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Vice-president of Shanghai Pulmonary Hospital,, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NALAN-01
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; 130-nm albumin-bound paclitaxel; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant PD-1 antibody puls chemotherapy (Experimental): Neoadjuvant treatment (PD-1 antibody+carboplatin+pemetrexed or nab-paclitaxel ) will start within 1-3 days from enrollment. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery. Before surgery a tumor assessment will be done. Patients with stable disease or partial response may be considered for surgery.
  Surgery: Surgery must be done within the 4rd-6th week from day 1 cycle 3 of neoadjuvant treatment (day 29-43 after day 1 of cycle 3) Adjuvant treatment: Patients that are R0 confirmed by surgical pathology evaluation will receive the first adjuvant administration within the 2rd to 8th week from surgery. Three cycles of combinded adjuvant treatment (PD-1 antibody+carboplatin+pemetrexed or nab-paclitaxel ) will be administered. Thirteen cycles of PD-1 antibody will start within day 21-24 days from day 1 of adjuvant cycle 2.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed or Nab-paclitaxel; Drug: PD-1 antibody
- Neoadjuvant chemotherapy (Active Comparator): Neoadjuvant treatment (carboplatin+pemetrexed or nab-paclitaxel ) will start within 1-3 days from enrollment/randomisation. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery. Before surgery a tumor assessment will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  Surgery: Surgery must be done within the 4rd-6th week from day 1 cycle 3 of neoadjuvant treatment (day 29-43 after day 1 of cycle 3).
  Adjuvant treatment: Patients that are R0 confirmed by surgical pathology evaluation will receive the first adjuvant administration within the 2rd to 8th week from surgery. Three cycles of adjuvant treatment (carboplatin+pemetrexed or nab-paclitaxel ) will be administered.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed or Nab-paclitaxel

INTERVENTIONS:
Drug: Carboplatin — (IV, Q3W)
Drug: Pemetrexed or Nab-paclitaxel — Pemetrexed (Nonsquamous NSCLC) or Nab-paclitaxel (Squamous NSCLC) (IV, Q3W)
Drug: PD-1 antibody — (IV, Q3W)
  Arms: Neoadjuvant PD-1 antibody puls chemotherapy

SUMMARY:
This is a randomized, open label study designed to evaluate the efficacy and safety of neoadjuvant PD-1 antibody plus chemotherapy followed by surgery in resectable stage IIIA-N2 non-small cell lung cancer.

DETAILED DESCRIPTION:
This is an open-label, randomised, two-arm, phase II, multi-centre clinical trial. The proposed study will evaluate the efficacy and safety of preoperative administration PD-1 antibody plus chemotherapy in patients resectable stage IIIA-N2 NSCLC. Data obtained in this study will provide valuable information for planning further phase III clinical trials of anti-PD-1 and other immunotherapies in NSCLC, both in the peri-operative and advanced disease setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females aged ≥18 years.
* Pathologically diagnosed of non-small cell lung cancer.
* Diagnosed as stage IIIA- N2.The diagnosis standard of N2 is as below: Pts with resectable stage IIIA-N2 NSCLC confirmed by mediastinoscopy or EBUS and PET/CT.
* Tumor should be considered resectable before study entry by a multidisciplinary team.
* ECOG (Performance status) 0-1.
* Screening laboratory values must meet the following criteria and should be obtained within 7 days prior to randomization.

  i. Neutrophils ≥ 1500×109/L ii. Platelets ≥ 100 x×109/L iii. Hemoglobin > 9.0 g/dL iv. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min v. AST/ALT ≤ 3 x ULN vi. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) vii. The patients need to have a forced expiratory volume (FEV1) ≥ 1.2 liters or >40% predicted value viii. INR/APTT within normal limits.
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before randomization.
* All sexually active men and women of childbearing potential must use an effective contraceptive method (two barrier methods or a barrier method plus a hormonal method) during the study treatment and for a period of at least 12 months following the last administration of trial drugs.
* Patient capable of proper therapeutic compliance and accessible for correct follow-up.
* Measurable or evaluable disease (according to RECIST 1.1 criteria).

Exclusion Criteria:

* All patients carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function. In case of doubt please contact trial team.
* Patients with other active malignancy requiring concurrent intervention and/or concurrent treatment with other investigational drugs or anti-cancer therapy.
* Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
* Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information.
* Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Patients with history of allergy to study drug components excipients.
* Women who are pregnant or in the period of breastfeeding.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
PFS at 24 months | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  The PFS is defined as the time from diagnosis to relapse, progression or death, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, School of Medicine, Tongji University
Locations (8):
- China (8):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Changzheng Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shuguang Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospita, Hangzhou, Zhejiang